CLINICAL TRIAL: NCT06604221
Title: The Impact of Resistance Exercise on Symptom Burden in Older Patients Undergoing Maintenance Hemodialysis
Brief Title: Resistance Exercise in Hemodialysis Patients
Acronym: REHDP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teng Zeng (Other)
Collaborators: Shengjing Hospital (Other)
Responsible Party: Sponsor-Investigator, Teng Zeng, Graduate student, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024148
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis
Keywords: resistance exercise; hemodialysis; older people
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance Exercise Intervention Group (Experimental): Resistance exercise intervention plan, developed through expert meetings and integrated review summaries, consists of 27 items including: participant preparation, team preparation, exercise prescription FITT-VP, process monitoring, discontinuation criteria, termination criteria, recovery methods, outcome measures, and special considerations.
  Interventions: Behavioral: Resistance exercise intervention; Behavioral: Routine care
- control group (Active Comparator): Routine care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Resistance exercise intervention — The exercise prescription, developed through expert meetings and integrated review summaries, consists of 27 items including: participant preparation, team preparation, exercise prescription FITT-VP, process monitoring, discontinuation criteria, termination criteria, recovery methods, outcome measures, and special considerations.
  Other Names: intra dialysis resistance exercise
  Arms: Resistance Exercise Intervention Group
Behavioral: Routine care — 1.Pre-dialysis Assessment:
  1. Vital Signs: Monitor blood pressure, heart rate, temperature.
  2. Access Care: Check the vascular access site for signs of infection and patency. 2.During Dialysis:
  （1）Monitoring: Continuous vital signs and machine settings monitoring. （2）Fluid Management: Control fluid removal based on pre-dialysis weight. 3.Post-dialysis Care:
  1. Observation: Monitor for complications like hypotension, cramps, or bleeding.
  2. Weight Check: Weigh post-dialysis to verify fluid removal. 4.Education and Support:
  （1）Diet: Educate on dietary restrictions (potassium, phosphorus, fluids). （2）Medications: Advise on medication adjustments. 5.Psychosocial Support:
  （1）Provide emotional support and counseling.
  Other Names: Routine care for hemodialysis

SUMMARY:
The goal of this clinical trial is to learn if an intradialytic resistance exercise intervention works to reduce the symptom burden in older maintenance hemodialysis patients. It will also learn about safety of the intradialytic resistance exercise intervention program. The main questions it aims to answer are:

1. Does intradialytic resistance exercise effectively improve the number, frequency, and severity of symptoms in older patients?
2. What adverse events may occur among older dialysis patients during exercise?

Researchers will compare older dialysis patients who undergo the intradialytic resistance exercise intervention with those receiving standard care to observe whether resistance exercise can improve symptom burden.

Participants will:

1. Take an intradialytic resistance exercise intervention program developed through joint decision-making by rehabilitation experts, dialysis center physicians, nurses, and patients, conducted three times a week for 20 minutes each session, over a duration of three months.
2. Visit the hospital a monthly for texts and examinations.
3. Keep a diary of the types and frequency of adverse events during and after the exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

Age 60 years and above Stable on dialysis for ≥3 months Able to walk independently, no physical disability, and muscle strength ≥ Grade III Capable of understanding and complying with the requirements of this study Voluntarily signed an informed consent form

Exclusion Criteria:

Severe cardiovascular, cerebrovascular, respiratory, or neurological diseases, or other conditions that impair physical ability to exercise Serious infections, bleeding, trauma, or other conditions affecting physical status within the last 3 months Severe mental disorders or cognitive impairments Abnormal blood pressure (pre-dialysis systolic pressure ≥180mmHg, diastolic pressure ≥100mmHg) Hemoglobin (Hb) < 90g/L, Albumin (Alb) ≤ 32g/L Participation in other exercise or pharmacological interventions in the past 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-03 (Estimated); Primary Completion 2025-01-03 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Dialysis Symptom Index | From enrollment to the end of treatment at 12 weeks
  Kidney failure-related symptoms were assessed every month using the dialysis symptom index (DSI), a previously validated questionnaire Through this questionnaire, patients indicated the presence of 30 symptoms in the past month, resulting in a total sum score for symptom number ranging from 0 to 30. Additionally, for each symptom present, patients rated symptom burden on a five-point Likert scale, ranging from one for "not at all" to five for "very much" burdensome. Absent symptoms were assigned a score of zero, resulting in an overall symptom burden score ranging from zero to 150, with higher scores indicating larger burden.

SECONDARY OUTCOMES:
30 Seconds Sit To Stand Test | From enrollment to the end of treatment at 12 weeks
  A chair with a hard seat whose floor-to-seat height was 48 cm was stabilized by placing it against a wall. After a researcher explained the requirements and precautions to the participant, the participant was asked to sit with his or her feet exactly flat on the ground and his or her upper limbs folded across his or her chest and then to stand up all the way and sit down again without using his or her arms. And the participant was asked to repeat as many of the sit-to-stand actions as possible in 30 seconds, and the maximum number completed was recorded.
  Higher scores mean a better outcome.
Short Physical Performance Battery | From enrollment to the end of treatment at 12 weeks
  (SPPB) which consists of 3 timed components: 1) a 4-meter usual pace walk, 2) a five-repetition chair stand without using one's arms, and 3) a progressive test of standing balance. Times from each component were scored from 0-4, with higher scores corresponding to better performance.
Number of participants with abnormal laboratory tests results | From enrollment to the end of treatment at 12 weeks
  blood urea, blood creatinine, dialysis adequacy (Kt/V), hemoglobin, neutrophil-to-lymphocyte ratio, serum albumin, standardized protein catabolic rate, C-reactive protein, inflammatory factors

IPD SHARING:
Plan to Share IPD: No
1. Privacy Concerns: To protect participant privacy and confidentiality, given the sensitive nature of the data.
  2. Research Integrity: To maintain the integrity of the research and prevent potential misuse of the data outside the specific study objectives.
  3. Personal Decision: To retain control over data usage and ensure adherence to ethical standards and research protocols established for this study.